CLINICAL TRIAL: NCT05257057
Title: Frequency of Endometrial Cancer Precursors Associated with Lynch Syndrome
Status: Completed | Type: Observational
Sponsor: WellSpan Health (Other)
Responsible Party: Principal Investigator, Eav Lim, Principal Investigator, WellSpan Health
Other Study IDs: 1403922-5
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2024-04

CONDITIONS: Lynch Syndrome; Endometrial Cancer; Endometrial Hyperplasia; Mismatch Repair Deficiency; Microsatellite Instability
Keywords: Lynch Syndrome; endometrial hyperplasia; endometrial cancer; immunohistochemistry; mismatch repair
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Endometrial Neoplasms; Endometrial Hyperplasia; Turcot syndrome; Microsatellite Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — No new biospecimens are retained. The biospecimens referenced are those that were already collected for tissue diagnosis of endometrial hyperplasia: endometrial biopsies, curettage specimens, and hysterectomy specimens. These are kept routinely in the pathology department on microscope slides post-procedure per hospital policy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Endometrial hyperplasia: These are patients with a diagnosis of endometrial hyperplasia at WellSpan in the study time frame diagnosed via endometrial biopsy, dilation and curettage, or hysterectomy.
  Interventions: Diagnostic Test: Immunohistochemical staining

INTERVENTIONS:
Diagnostic Test: Immunohistochemical staining — Immunohistochemistry will be performed on the endometrial tissue specimens

SUMMARY:
Given that there is a significant prevalence of Lynch syndrome among patients with endometrial cancer (about 5% of patients with endometrial cancer), and given there is a known risk of endometrial cancer among patients with endometrial hyperplasia (40% risk of pre-existing occult cancer with endometrial intraepithelial neoplasia), it is hypothesized that a diagnosis of endometrial hyperplasia may herald on-going risk of harboring a Lynch Syndrome gene mutation.

The purpose of this study is to examine endometrial hyperplasia specimens and compare the frequency of Lynch Syndrome gene mutations between endometrial hyperplasia and endometrial cancer subjects. This will provide a rationale and opportunity for earlier screening, and reduce colon cancer morbidity and mortality secondary to the Lynch syndrome gene.

DETAILED DESCRIPTION:
This is an observational cohort study. Tissue specimens obtained that have been labeled with the diagnosis of endometrial hyperplasia will be identified and their chart reviewed for demographic date of age, race, body mass index, and co-morbidities. The specimen will then be tested via immunohistochemistry for the mismatch repair proteins MLH1, PMS2, MSH2, or MSH 6. Their absence is indicative of Lynch Syndrome. Statistical analysis will then be performed to compare the incidence of Lynch syndrome in endometrial hyperplasia with Lynch Syndrome in endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Appropriate specimen, hysterectomy or biopsy with final labeled diagnosis of endometrial hyperplasia of any grade

Exclusion Criteria:

* Any specimen that is later associated with endometrial cancer in subsequent pathology exam

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who underwent tissue sampling of any type and received a pathologic diagnosis of endometrial hyperplasia at WellSpan from 2014-2022.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2019-05-08 (Actual); Primary Completion 2023-06-02 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Lynch Syndrome Screen Positive Rate | 2014-2022
  This is the rate of subjects who screen positive for Lynch Syndrome based on immunohistochemical staining

CONTACTS AND LOCATIONS:
Overall Officials: Eav Lim, DO, Principal Investigator — WellSpan Health-York Cancer Center
Locations (1):
- WellSpan, York, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hampel H, de la Chapelle A. The search for unaffected individuals with Lynch syndrome: do the ends justify the means? Cancer Prev Res (Phila). 2011 Jan;4(1):1-5. doi: 10.1158/1940-6207.CAPR-10-0345. PMID 21205737
- [Background] Sehgal R, Sheahan K, O'Connell PR, Hanly AM, Martin ST, Winter DC. Lynch syndrome: an updated review. Genes (Basel). 2014 Jun 27;5(3):497-507. doi: 10.3390/genes5030497. PMID 24978665
- [Background] Ryan NAJ, Blake D, Cabrera-Dandy M, Glaire MA, Evans DG, Crosbie EJ. The prevalence of Lynch syndrome in women with endometrial cancer: a systematic review protocol. Syst Rev. 2018 Aug 16;7(1):121. doi: 10.1186/s13643-018-0792-8. PMID 30115102
- [Background] Wang Y, Wang Y, Li J, Cragun J, Hatch K, Chambers SK, Zheng W. Lynch syndrome related endometrial cancer: clinical significance beyond the endometrium. J Hematol Oncol. 2013 Mar 25;6:22. doi: 10.1186/1756-8722-6-22. PMID 23531335
- [Background] ACOG Practice Bulletin No. 147: Lynch syndrome. Obstet Gynecol. 2014 Nov;124(5):1042-1054. doi: 10.1097/01.AOG.0000456325.50739.72. No abstract available. PMID 25437740
- [Background] Kurman RJ, Kaminski PF, Norris HJ. The behavior of endometrial hyperplasia. A long-term study of "untreated" hyperplasia in 170 patients. Cancer. 1985 Jul 15;56(2):403-12. doi: 10.1002/1097-0142(19850715)56:23.0.co;2-x. PMID 4005805
- [Background] de Leeuw WJ, Dierssen J, Vasen HF, Wijnen JT, Kenter GG, Meijers-Heijboer H, Brocker-Vriends A, Stormorken A, Moller P, Menko F, Cornelisse CJ, Morreau H. Prediction of a mismatch repair gene defect by microsatellite instability and immunohistochemical analysis in endometrial tumours from HNPCC patients. J Pathol. 2000 Nov;192(3):328-35. doi: 10.1002/1096-9896(2000)9999:99993.0.CO;2-2. PMID 11054716
- [Background] Han SJ, Kim MK. Clinical significance of mismatch repair genes immunohistochemical expression of complex endometrial hyperplasia. Obstet Gynecol Sci. 2015 Mar;58(2):106-11. doi: 10.5468/ogs.2015.58.2.106. Epub 2015 Mar 16. PMID 25798423
- [Background] Horn LC, Meinel A, Handzel R, Einenkel J. Histopathology of endometrial hyperplasia and endometrial carcinoma: an update. Ann Diagn Pathol. 2007 Aug;11(4):297-311. doi: 10.1016/j.anndiagpath.2007.05.002. PMID 17630117
- [Background] Huang M, Djordjevic B, Yates MS, Urbauer D, Sun C, Burzawa J, Daniels M, Westin SN, Broaddus R, Lu K. Molecular pathogenesis of endometrial cancers in patients with Lynch syndrome. Cancer. 2013 Aug 15;119(16):3027-33. doi: 10.1002/cncr.28152. Epub 2013 Jun 12. PMID 23760948
- [Background] Ichikawa Y, Tsunoda H, Takano K, Oki A, Yoshikawa H. Microsatellite instability and immunohistochemical analysis of MLH1 and MSH2 in normal endometrium, endometrial hyperplasia and endometrial cancer from a hereditary nonpolyposis colorectal cancer patient. Jpn J Clin Oncol. 2002 Mar;32(3):110-2. doi: 10.1093/jjco/hyf026. PMID 11956307
- [Background] Ketabi Z, Gerdes AM, Mosgaard B, Ladelund S, Bernstein I. The results of gynecologic surveillance in families with hereditary nonpolyposis colorectal cancer. Gynecol Oncol. 2014 Jun;133(3):526-30. doi: 10.1016/j.ygyno.2014.03.012. Epub 2014 Mar 13. PMID 24631699
- [Background] Manchanda R, Saridogan E, Abdelraheim A, Johnson M, Rosenthal AN, Benjamin E, Brunell C, Side L, Gessler S, Jacobs I, Menon U. Annual outpatient hysteroscopy and endometrial sampling (OHES) in HNPCC/Lynch syndrome (LS). Arch Gynecol Obstet. 2012 Dec;286(6):1555-62. doi: 10.1007/s00404-012-2492-2. Epub 2012 Aug 4. PMID 22865035
- [Background] Sutter C, Dallenbach-Hellweg G, Schmidt D, Baehring J, Bielau S, von Knebel Doeberitz M, Gebert J. Molecular analysis of endometrial hyperplasia in HNPCC-suspicious patients may predict progression to endometrial carcinoma. Int J Gynecol Pathol. 2004 Jan;23(1):18-25. doi: 10.1097/01.pgp.0000101085.35393.4a. PMID 14668545
- [Background] Vierkoetter KR, Kagami LA, Ahn HJ, Shimizu DM, Terada KY. Loss of Mismatch Repair Protein Expression in Unselected Endometrial Adenocarcinoma Precursor Lesions. Int J Gynecol Cancer. 2016 Feb;26(2):228-32. doi: 10.1097/IGC.0000000000000606. PMID 26807560